CLINICAL TRIAL: NCT03582956
Title: Effect of Adiposity on Hepatic and Peripheral Insulin Resistance in Type 1 Diabetes
Acronym: T1D
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2000023149; 1K23DK115894-01A1 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-07-11 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Type1 Diabetes Mellitus; Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Adolescent Overweight (Other): Adolescents with T1D and overweight/obesity
  Interventions: Procedure: Euglycemic hyperinsulinemic clamp with tracer enhancement
- Adolescent Typical (Other): Lean adolescents with T1D
  Interventions: Procedure: Euglycemic hyperinsulinemic clamp with tracer enhancement
- Young Adult (Other): Young adults with T1D with a euglycemic hyperinsulinemic clamp with tracer enhancement
  Interventions: Procedure: Euglycemic hyperinsulinemic clamp with tracer enhancement

INTERVENTIONS:
Procedure: Euglycemic hyperinsulinemic clamp with tracer enhancement — To characterize the impact of adiposity on metabolism during puberty, adolescents will undergo the euglycemic hyperinsulinemic clamp study with tracer enhancement.
  Arms: Adolescent Overweight; Adolescent Typical
Procedure: Euglycemic hyperinsulinemic clamp with tracer enhancement — A comparison control group of 36 lean young adults with T1D will also be enrolled, since they will be unaffected by the adverse metabolic effects of puberty or obesity.
  Arms: Young Adult

SUMMARY:
The purpose of this study is to assess the effects of adiposity on resistance to insulin's ability to suppress hepatic glucose production and to stimulate peripheral glucose metabolism in adolescents with type 1 diabetes. In addition, this study will also examine the role of fatty liver disease on the insulin resistance of obesity in adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
A major focus of this program of research will be directed at advancing the understanding of the metabolic consequences of obesity and puberty in adolescents with T1D. Thus, an innovative aspect of this research is that it will be the first to use these sophisticated metabolic techniques to examine the effects of obesity and hepatic steatosis on insulin sensitivity in pubertal adolescents with T1D; namely, the 2-step hyperinsulinemic euglycemic clamp with tracer enhancement, which will allow for definition of hepatic and peripheral insulin resistance, glycerol turnover, and glucose and fat oxidation. Further, a second novel aspect is that this will be the first study to utilize gold standard MRI methods to quantify and compare intrahepatic fat content in lean and obese adolescents with T1D. This will allow a global and more detailed understanding of the potential alterations of insulin's effects on key insulin sensitive tissues in youth that are impacted by both T1D and obesity. Furthermore, evaluation of biomarkers for insulin resistance and fatty liver disease in this population will be performed for the first time.

ELIGIBILITY:
Inclusion Criteria:

* All Participants:

  1. Clinical diagnosis of T1D
  2. HbA1c ≤9%
  3. Diabetes duration of at least 12 months

Adolescents with T1D:

1. Age 12-16 years
2. BMI <75th for lean pediatric subjects, > 85th percentile for overweight/obese pediatric subjects;
3. Tanner stage 2-5
4. Parent able to provide written consent and participant able to provide assent
5. Not meeting MRI safety criteria
6. Claustrophobia that will prevent participation in the MRI

Lean, young adults with T1D:

1. Age 18-24 years
2. BMI 18.5-24.9 kg/m2
3. Able to provide written consent.

Exclusion Criteria:

1. Use of adjunctive diabetes medications
2. Weight loss medications within the past six months
3. Current psychiatric disorders, including eating disorders (DSM-V criteria)
4. Known liver disease other than nonalcoholic hepatic steatosis
5. Females who are pregnant or lactating
6. Anemia or another medical condition that precludes participation in the study

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Van Name, MD, Principal Investigator — Yale University
Locations (1):
- Yale Pediatric Diabetes Research Program, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant enrolled but did not have any baseline or study data obtained due to scheduling conflicts.
Groups:
- Adolescent Overweight: Adolescents with T1D and body mass index ≥85% will undergo a euglycemic hyperinsulinemic clamp with tracer enhancement.
  Euglycemic hyperinsulinemic clamp with tracer enhancement: To characterize the impact of adiposity on metabolism during puberty, adolescents will undergo the euglycemic hyperinsulinemic clamp study with tracer enhancement.
- Adolescent Typical: Adolescents with T1D and body mass index <75% will undergo a euglycemic hyperinsulinemic clamp with tracer enhancement.
  Euglycemic hyperinsulinemic clamp with tracer enhancement: To characterize the impact of adiposity on metabolism during puberty, adolescents will undergo the euglycemic hyperinsulinemic clamp study with tracer enhancement.
- Young Adult: Young Adults with T1D and body mass index 18.5 to <25 kg/m2 will undergo a euglycemic hyperinsulinemic clamp with tracer enhancement.
Period: Overall Study
Arm/Group | Adolescent Overweight | Adolescent Typical | Young Adult
Started | 13 | 7 | 2
Completed | 13 | 7 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for each group.
Groups:
- Adolescent Typical Weight: Adolescents with T1D and body mass index <75% will undergo a euglycemic hyperinsulinemic clamp with tracer enhancement.
  Euglycemic hyperinsulinemic clamp with tracer enhancement: To characterize the impact of adiposity on metabolism during puberty, adolescents will undergo the euglycemic hyperinsulinemic clamp study with tracer enhancement.
- Adolescent Overweight/Obese: Adolescents with T1D and body mass index ≥85% will undergo a euglycemic hyperinsulinemic clamp with tracer enhancement.
  Euglycemic hyperinsulinemic clamp with tracer enhancement: To characterize the impact of adiposity on metabolism during puberty, adolescents will undergo the euglycemic hyperinsulinemic clamp study with tracer enhancement.
- Total: Total of all reporting groups
Arm/Group | Adolescent Typical Weight | Adolescent Overweight/Obese | Young Adult | Total
Number analyzed (Participants) | 7 | 13 | 2 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.11) | 14.5 (1.19) | 20.65 (2.48) | 15.57 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 0 | 12
  Male | 3 | 5 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 6 | 11 | 2 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 11 | 2 | 20
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 13 | 2 | 22
percentage of glycated hemoglobin [Mean (Standard Deviation); unit: percentage] | 7.32 (0.60) | 7.74 (0.41) | 6.35 (0.49) | 7.48 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Glucose Metabolism
Description: Insulin function will be measured using a euglycemic hyperinsulinemic clamp procedure. A clamp measures insulin sensitivity. During the low does insulin phase, this reflects hepatic glucose metabolism, which is reported here. A higher glucose infusion rate number indicates more sensitivity to insulin; a lower number means more resistance to insulin.
Time Frame: 120 minutes
Population: Only adolescents were analyzed due to the availability of data in the aftermath of the COVID shutdown- data were not collected on the young adult group.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Adolescent Overweight | Adolescent Typical
Number analyzed (Participants) | 12 | 7
mg/kg/min | 1.74 (0.77) | 1.56 (0.41)
Statistical Analysis 1: Comparison: Adolescent Overweight vs Adolescent Typical; Test type: Superiority; p = 0.525, t-test, 2 sided

2. Primary Outcome: Rate of Lipid Metabolism
Description: Insulin function will be measured using a euglycemic hyperinsulinemic clamp procedure. A clamp measures insulin sensitivity. During the low dose insulin phase, glycerol turnover (rate of appearance) can reflect adipose specific insulin sensitivity, which is reported here. Insulin should suppress glycerol turnover. A higher number reflects more resistance to insulin; a lower number means more sensitivity to insulin.
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Adolescent Overweight | Adolescent Typical
Number analyzed (Participants) | 12 | 7
mg/kg/min | 0.099 (0.077) | 0.12 (0.099)
Statistical Analysis 1: Comparison: Adolescent Overweight vs Adolescent Typical; Test type: Superiority; p = 0.607, t-test, 2 sided

3. Primary Outcome: Hepatic Sensitivity to Low Dose Insulin
Description: Insulin function will be measured using a euglycemic hyperinsulinemic clamp procedure. A clamp measures insulin sensitivity. Insulin should suppress glucose production. Change of the glucose rate of appearance (which is reported here, and the glucose rate of appearance is measured here utilizing isotopic enrichment) during the low dose insulin phase reflects hepatic sensitivity to insulin. A greater degree of decline reflects more sensitivity to insulin; a smaller number means more resistance to insulin.
  This is calculated as the low dose insulin phase glucose rate of appearance minus the baseline phase glucose rate of appearance, divided by the basal phase glucose rate of appearance and multiplied x 100.
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of suppression of Ra glucose
Arm/Group | Adolescent Overweight | Adolescent Typical
Number analyzed (Participants) | 12 | 7
percentage of suppression of Ra glucose | -27.9 (25.8) | -35.8 (15.3)
Statistical Analysis 1: Comparison: Adolescent Overweight vs Adolescent Typical; Test type: Superiority; p = 0.466, t-test, 2 sided

4. Primary Outcome: Peripheral Sensitivity to High Dose Insulin
Description: Insulin function will be measured using a euglycemic hyperinsulinemic clamp procedure. A clamp measures insulin sensitivity. Insulin should suppress glucose production. Change of the glucose rate of appearance (which is reported here, and the glucose rate of appearance is measured here utilizing isotopic enrichment) during the high dose phase reflects peripheral sensitivity to insulin. A greater degree of decline reflects more sensitivity to insulin; a smaller number means more resistance to insulin.
  This is calculated as the high dose insulin phase glucose rate of appearance minus the baseline phase glucose rate of appearance, divided by the basal phase glucose rate of appearance and multiplied x 100.
Time Frame: 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of suppression of Ra glucose
Arm/Group | Adolescent Overweight | Adolescent Typical
Number analyzed (Participants) | 11 | 7
percentage of suppression of Ra glucose | -75.99 (58.8) | -96.48 (32.5)
Statistical Analysis 1: Comparison: Adolescent Overweight vs Adolescent Typical; Test type: Superiority; p = 0.414, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 hours
Description: This is not a longitudinal study, and there was no intervention
Groups:
- Adolescent Overweight: The study aims to enroll 36 adolescents with T1D and overweight/obesity, 36 lean adolescents with T1D, and 36 young adults with T1D that will receive a euglycemic hyperinsulinemic clamp with tracer enhancement.
  Euglycemic hyperinsulinemic clamp with tracer enhancement: To characterize the impact of adiposity on metabolism during puberty, adolescents will undergo the euglycemic hyperinsulinemic clamp study with tracer enhancement.
- Adolescent Typical: The study aims to enroll 36 adolescents with T1D and overweight/obesity, 36 lean adolescents with T1D, and 36 young adults with T1D a euglycemic hyperinsulinemic clamp with tracer enhancement.
  Euglycemic hyperinsulinemic clamp with tracer enhancement: To characterize the impact of adiposity on metabolism during puberty, adolescents will undergo the euglycemic hyperinsulinemic clamp study with tracer enhancement.
- Young Adult: Young adults with T1D a euglycemic hyperinsulinemic clamp with tracer enhancement.
Arm/Group | Adolescent Overweight | Adolescent Typical | Young Adult
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03582956/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03582956/ICF_001.pdf